CLINICAL TRIAL: NCT07102433
Title: CHESS - Complexity and Outcomes in Health, Education, and Social Support Among Children and Young People With Life-limiting Conditions: Establishing a Multisectoral Collaboration and Conceptual Framework to Advance Evidence and Practice.
Brief Title: Complexity in Health, Education, and Social Support for Children and Young People With Life-limiting Conditions.
Acronym: CHESS
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRAS 356844; NIHR207608 (Other: National Institute for Health and Care Research)
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-07

CONDITIONS: Complex Care; Medical Complexity; Pediatrics; Life-limiting Illness; Life-threatening Illness
Keywords: Medical complexity; Pediatric palliative care; Life-limiting conditions; Life-threatening conditions; Children and young people
MeSH Terms: interventions — Caregivers; Educational Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interview and Workshop Participants: Interview and workshop participants will be formed from the following inclusion criteria:
  Children and Young People (CYP):
  * Aged 5-17 years
  * Diagnosed with a life-limiting condition (as defined by Together for Short Lives)
  Parents/Carers:
  * Parent/carer of a child aged 0-17 years with a life-limiting condition
  * Bereaved parent, where bereavement occurred ≥3 months ago
  Professionals (Health, Social Care, Education):
  * Working with CYP with life-limiting conditions for at least 6 months
  * Includes medical, nursing, allied health, social care, and educational professionals
  Workshop Participants:
  * Any of the above stakeholder types
  * Must be able to provide informed consent or assent
  Interventions: Other: Children and young people with life-limiting conditions, their parents/carers, and professionals across healthcare, education, and social care sectors.

INTERVENTIONS:
Other: Children and young people with life-limiting conditions, their parents/carers, and professionals across healthcare, education, and social care sectors. — Children and young people with life-limiting conditions, their parents/carers, and professionals across healthcare, education, and social care sectors.

SUMMARY:
Children and young people (CYP) with life-limiting conditions represent a growing population with complex care needs that span health, education, and social care systems. These children often have multiple diagnoses, rely on medical technologies, and experience prolonged trajectories of illness. Despite this, care remains fragmented, services are poorly integrated, and definitions of "complexity" are variable, inconsistent, and inadequately reflect the lived experience of families and the perspectives of professionals.

The CHESS (Complexity in Health, Education, and Social Support) study aims to develop a shared, evidence-informed understanding of "complexity" in the context of CYP with life-limiting conditions. The study will be delivered by a multi-disciplinary, multisectoral research team and is funded by a National Institute for Health and Care Research (NIHR) Programme Development Grant. This research will provide the foundational work to inform the design and implementation of a future NIHR Programme Grant focused on the development and testing of a child-centred, nationally applicable case mix classification system to support integrated multisector care and resource allocation.

This qualitative study involves two stages. Stage 1 consists of semi-structured interviews with (i) CYP aged 5-17 years with a life-limiting condition, (ii) parents/carers (including bereaved parents and parents of children aged under 5 years), and (iii) professionals across healthcare, social care, and education sectors. These interviews aim to elicit stakeholder understandings of "complexity," how it is experienced and enacted in care, and the implications for service access, coordination, and outcomes.

Stage 2 comprises a series of stakeholder workshops to review, refine, and synthesise findings from Stage 1 and a parallel realist review. Using consensus methods including the Nominal Group Technique, the workshops will co-develop a cross-sectoral conceptual definition of "complexity" and produce a logic model to guide integrated care delivery for this population.

The CHESS study seeks to address a critical evidence gap in how complexity is understood, measured, and supported across systems. By incorporating the voices of children, families, and professionals across sectors, this study will generate new conceptual clarity, build a foundation for improved outcomes, and contribute directly to the national agenda on equity, quality, and integration in paediatric palliative and complex care.

DETAILED DESCRIPTION:
1. Background and Rationale

   Children and young people living with life-limiting conditions (LLCs) represent a population with profoundly complex and multidimensional needs. These conditions, which include both life-limiting and life-threatening diagnoses, are characterised by an absence of curative options and, in many cases, uncertain illness trajectories. Advances in medical care mean that children often survive longer than previously expected, but with increasing medical, social, and educational complexity.

   Care for this group typically spans multiple sectors: highly specialised medical teams, allied health professionals, children's hospices, social services, and educational systems. Parents frequently report fragmented services, difficulties in navigating between health, education, and social care, and inequitable access to essential resources such as medical technologies, equipment, and tailored educational support. Despite being a relatively small population, these children account for disproportionately high resource utilisation, including frequent and prolonged hospital admissions, intensive care stays, and substantial reliance on community-based services.

   The absence of a shared definition of "complexity" across health, education, and social care settings poses a major barrier to effective care delivery. Services lack a consistent framework for recognising, measuring, and responding to complexity, resulting in inequitable distribution of resources and difficulties in evaluating outcomes. Research into children with neurodisability has attempted to capture aspects of complexity, but such tools are impractical in routine settings and insufficiently inclusive of the breadth of needs among children with LLCs.

   Previous initiatives have shown progress in developing outcome measures in paediatric palliative care and in mapping models of end-of-life care. However, no work has systematically brought together children, families, professionals, and policy stakeholders across sectors to build a conceptual model of complexity. In contrast, adult palliative care in the UK has successfully developed and implemented classification frameworks that inform both care and policy. A similar evidence base is urgently needed for children.

   The CHESS study (Complexity in Health, Education, and Social Support) addresses this evidence gap. By drawing on interviews with children, parents, and professionals, and by convening cross-sector workshops, this study will generate a consensus definition of complexity and a logic model of integrated multisector care. This framework will inform the development of a child-centred, nationally applicable classification system for future research and service planning.
2. Study Purpose and Objectives

   The overarching purpose of CHESS is to build an evidence-based conceptual model of complexity in children with LLCs that is recognised across health, education, and social care sectors. This study is funded by the UK National Institute for Health and Care Research (NIHR) through a Programme Development Grant, and its outputs will underpin a future Programme Grant to design and test a case-mix classification for integrated care.

   Primary Objective

   To develop a cross-sector, evidence-based conceptual model of complexity for children with LLCs, derived from qualitative interviews and stakeholder workshops.

   Stage 1: Interviews

   To capture the perspectives of children, parents (including bereaved parents), and professionals on the meaning and operationalisation of "complexity."

   To understand children's experiences of their care needs, the supports they value, and barriers to meeting these needs.

   To identify parents' views on gaps in provision and how complexity influences the challenges they face.

   To explore professionals' definitions of complexity and their approaches to care planning.

   Stage 2: Workshops

   To build consensus on how complexity is defined and operationalised across sectors.

   To identify key components, processes, and outcomes essential for delivering integrated care.

   To develop a logic model of integrated care, with agreed indicators and outputs that reflect complexity.

   Secondary Objectives

   To establish a collaborative research partnership across multiple disciplines and sectors.

   To generate findings that support equitable resource allocation and guide future policy.

   To strengthen patient and public involvement (PPI) in conceptualising and shaping research on complexity.
3. Study Design and Methodology

   This is a qualitative, multi-stage study consisting of two sequential components:

   Stage 1 - Semi-structured Interviews

   Participants: children (aged 5-17 years), parents/carers (including bereaved parents and parents of children aged under 5), and professionals (health, social care, education).

   Purpose: to capture diverse views on complexity, using purposive sampling to ensure variation in age, condition, ethnicity, socio-economic status, and professional background.

   Method: in-depth, semi-structured interviews, supported by age-appropriate tools (e.g., Talking Mats™, draw/play methods).

   Stage 2 - Stakeholder Workshops

   Three initial workshops (~30 participants each) involving parents, professionals, researchers, and carers.

   A final consensus workshop (~30 participants) using Nominal Group Technique to refine definitions and logic models.

   Data: transcripts and facilitated discussions analysed to develop a consensus definition and a framework for integrated care.

   The design is informed by a pragmatist research paradigm, acknowledging the experiential and contextual nature of complexity. Appreciative Inquiry principles will guide workshops, focusing on "what works" in integrated care.

   Study Duration: 9 months 31 days.
4. Participants: Eligibility and Recruitment 4.1 Children and Young People

   Inclusion

   Aged 5-17 years.

   Diagnosed with a life-limiting condition (as defined by Together for Short Lives).

   Able to communicate verbally, through play/drawing, Talking Mats™, or via a parent proxy.

   Exclusion

   Unable to communicate using available methods.

   Non-English speakers where NHS translation services are unavailable.

   Considered by clinical staff at participating centres to be at risk of undue distress.

   Recruitment

   Through NHS trusts, hospices, and community organisations serving children with LLCs.

   Care teams identify eligible children and seek parental consent for contact.

   4.2 Parents and Carers

   Inclusion

   Parents/carers of children aged 0-17 years with an LLC.

   Bereaved parents (>3 months since bereavement).

   Exclusion

   Recently bereaved (<3 months).

   Unable to provide informed consent.

   At risk of psychological harm if participating.

   4.3 Professionals

   Inclusion

   Healthcare (medicine, nursing, allied health), social care, or education professionals with ≥6 months' experience caring for children with LLCs.

   Exclusion

   Professionals with <6 months' experience.

   4.4 Workshop Participants

   Drawn from interview participants and wider networks.

   Must be able to provide informed consent.

   Children are not included in workshops.

   Sample Size Estimates

   Interviews: 10-20 children, ≥30 parents/carers, ≥30 professionals.

   Workshops: ~90 participants across three initial workshops and one consensus session.
5. Study Procedures 5.1 Interviews

   Conducted face-to-face or via secure video (Microsoft Teams).

   Duration: children (30-60 min), parents (60-90 min), professionals (~60 min).

   Interviews will be audio-recorded, transcribed verbatim, pseudonymised.

   Children's interviews will include rapport-building, discussion of daily life, care needs, support experiences, and hopes for improvement.

   Parents will be asked about daily care, experiences with services, barriers, and views on complexity.

   Professionals will discuss definitions of complexity, service challenges, and approaches to integration.

   Participants will receive £20 vouchers and reimbursement for travel/childcare.

   5.2 Workshops

   Conducted remotely via Microsoft Teams to maximise accessibility.

   Three initial workshops will generate broad definitions and frameworks.

   A final workshop will synthesise findings using Nominal Group Technique.

   Outputs: consensus definition of complexity and a preliminary logic model.
6. Data Management and Analysis Plan

   All identifiable data (e.g., consent forms, audio/video files) will be stored separately from transcripts.

   Data will be held on secure, password-protected King's College London SharePoint servers.

   Audio files will be transcribed by a GDPR-compliant service; audio destroyed after transcription.

   Video recordings of Talking Mats™ sessions will be analysed then deleted.

   Interview data will be analysed using Framework Analysis, ensuring transparency, coding consistency, and traceability.

   Workshop data will be analysed using Nominal Group Technique and the CDC guide for developing logic models.

   Emergent findings will be triangulated across children, parents, and professionals.
7. Statistical Considerations

   This is a qualitative study; no hypothesis testing or quantitative statistical modelling is planned. Sample sizes are based on principles of pragmatic saturation, ensuring adequate diversity and depth of data.

   Interviews: expected saturation with ~60-80 participants.

   Workshops: sufficient numbers to capture balance between parents and professionals, with consensus tested through structured group methods.
8. Ethics, Safety, and Risk Management

   Ethical Review: The study requires NHS REC and HRA approval.

   Informed Consent/Assent

   Parents provide written consent for themselves and for children under 16.

   Children aged 5-15 provide assent; those aged 16-17 provide consent where capacity is confirmed.

   Bereaved parents must be at least 3 months post-bereavement.

   Managing Distress

   Researchers trained in qualitative methods for sensitive topics.

   Distress protocol includes pausing/stopping interviews, signposting to support, and notifying care teams if needed.

   No disclosure of prognosis or new medical information will occur during interviews.

   Adverse Events

   Although AEs and SAEs are unlikely in qualitative research, any unexpected events (e.g., acute distress) will be recorded and reported according to NIHR and sponsor policies.

   Safeguarding

   The study complies with NIHR and KCL safeguarding guidelines.

   Children may have a parent or trusted adult present during interviews.
9. Oversight, Roles, and Responsibilities

   Sponsor: King's College London - responsible for study initiation, management, and monitoring.

   Funder: NIHR Programme Development Grant (NIHR207608).

   Chief Investigator: Prof. Richard Harding (Cicely Saunders Institute).

   Co-Investigators: Multidisciplinary team spanning paediatric medicine, social care, ethics, education, and patient/public representation.

   Steering Committee: Includes patient and public involvement (PPI) members and professionals, meeting monthly to guide recruitment, methodology, and interpretation.

   Auditing/Monitoring: Sponsor may audit per UK Policy Framework for Health and Social Care.
10. Dissemination and Impact

Findings will inform the development of a cross-sector conceptual model of complexity, which will underpin a subsequent NIHR Programme Grant proposal. Dissemination plans include:

Peer-reviewed publications in palliative care, paediatrics, education, and social policy journals.

Presentations at international conferences.

A public launch of the consensus definition, involving parents and carers.

Sharing findings with NHS England, local authorities, and professional associations.

Lay summaries and online dissemination co-developed with PPI representatives.

Ultimately, the study aims to provide a nationally applicable, child-centred framework for understanding complexity in LLCs, enabling more equitable service design, evaluation, and resource allocation.

ELIGIBILITY:
Stage 1 - Interviews

Inclusion Criteria:

* Children (5-17 years) with any life-limiting condition defined using the UK Together for Short Lives widely adopted 4 categories of life-limiting/life-threatening conditions among children.
* Parents/carers of children (0-17 years old) with a life-limiting conditions.
* Bereaved parents of a child who had a life-limiting condition (at least 3 months since bereavement).
* Healthcare professionals (medicine, nursing, allied health professionals), social care providers, education teaching and therapy staff with > 6 months experience of caring for children with life-limiting conditions.

Exclusion Criteria:

* Children unable to communicate via an interview, using 'draw and talk' or play methods, Talking MatsTM, or via their parents.
* Children that speak languages not supported by NHS translation services.
* Any child or young person for whom the PI believes participation in the study may induce undue psychological distress.
* Parents/carers are unable to provide consent/assent to participate in interviews.
* Parents/carers that speak languages not supported by NHS translation services.
* Parents who are recently bereaved (<3 months).
* Any parent/carer for whom the PI believes participation in the study may induce undue psychological distress (e.g. parents of children who may be receiving end-of-life care).
* Professionals with <6 months experience of caring for children with life-limiting conditions.

Stage 2 - Workshops

Inclusion criteria:

* Parents or carers of children with a life-limiting condition (0-17 years old).
* Bereaved parents of a child who had a life-limiting condition (at least 3 months since bereavement).
* Researchers working with or in the field of complexity in children with life-limiting conditions.
* Professionals across child health, social care, and education with experience of working with children with life-limiting conditions for >6 months.

Exclusion criteria:

* Professionals across child health, social care, and education with <6 months of experience working with children with life-limiting conditions.
* Parents, carers, or professionals that are unable to provide consent or assent.
* Children with life-limiting/life-threatening conditions will not be included in the workshops
* Parents who are recently bereaved (<3 months) of a child who had a life-limiting condition.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises: (1) children and young people aged 5-17 years with a life-limiting condition; (2) parents or carers of children aged 0-17, including bereaved parents (≥3 months post-bereavement); and (3) professionals from health, education, and social care with ≥6 months' experience supporting this population. Participants will be recruited from five NHS and hospice sites across England, selected for variation in geography, population served, and service model. Purposive sampling will be used to ensure diversity in age, diagnosis, ethnicity, socioeconomic status, and care setting. Professionals will be drawn from a range of disciplines across sectors using our professional networks.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Study Objective | Total Duration of study - August 2025 to July 2026.
  Use findings from stakeholder interviews and workshops to develop a cross-sector evidence-based conceptual model of complexity to inform delivery and assessment of high quality and integrated care.
Interviews - Research Question | Total study duration - August 2025 to July 2026
  What does 'complexity' mean to stakeholders in relation to children with life-limiting conditions, with respect to their health, social care, and educational needs and how they are understood, planned, and delivered?
Workshops Research Questions | Total study duration - August 2025 to July 2026
  1. How is 'complexity' defined and operationalised across health, social care, and education for children and young people with life-limiting conditions?
  2. What components and processes are important for the delivery of integrated complex care?
  3. What outputs and indicators signal 'complexity' and appropriate care delivery?
  4. Which processes and outcomes are meaningful to evaluate?

CONTACTS AND LOCATIONS:
Overall Officials: Fliss Murtagh, Principal Investigator — Hull York Medical School; Mary Baginsky, Principal Investigator — King's College London; Diane Sellers, Principal Investigator — Chailey Clinical Services, Sussex Community NHS Foundation Trust; Lucy Coombes, Principal Investigator — Royal Marsden NHS Foundation Trust; Mary Salama, Principal Investigator — Birmingham Children's Hospital; Bobbie Farsides, Principal Investigator — Brighton and Sussex Medical School; Gabriella L Walker, Principal Investigator — Patient and Public Representative; Pru Holder, Principal Investigator — King's College London; Abinaya Chandrasekar, Principal Investigator — King's College London
Locations (5):
- United Kingdom (5):
  - Birmingham Children's Hospital, Birmingham
  - Chailey Clinical Services, Sussex Community NHS Foundation Trust, Chailey
  - Shooting Star Children's Hospices, Hampton
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: No
This is a qualitative study involving in-depth interviews and stakeholder workshops with children, parents (including bereaved parents), and professionals. Due to the nature of the data collected-highly personal, context-specific, and potentially identifiable-even after de-identification, individual participant data (IPD) will not be shared publicly. This decision is guided by ethical considerations, the sensitivity of participant narratives, and the need to preserve confidentiality in accordance with informed consent agreements and data governance policies. Summarised findings will be shared through academic publications, public reports, and stakeholder events.

REFERENCES:
- [Background] Rahimzadeh V, Bartlett G, Longo C, Crimi L, Macdonald ME, Jabado N, Ells C. Promoting an ethic of engagement in pediatric palliative care research. BMC Palliat Care. 2015 Oct 16;14:50. doi: 10.1186/s12904-015-0048-5. PMID 26474573
- [Background] Low, J. (2019). A pragmatic definition of the concept of theoretical saturation. Sociological Focus 52(2), 131-139.
- [Background] Fields D, Fraser LK, Taylor J, Hackett J. What does 'good' palliative care look like for children and young people? A qualitative study of parents' experiences and perspectives. Palliat Med. 2023 Mar;37(3):355-371. doi: 10.1177/02692163231154300. Epub 2023 Feb 24. PMID 36825577
- [Background] Fisher V, Atkin K, Fraser LK. The health of mothers of children with a life-limiting condition: A qualitative interview study. Palliat Med. 2022 Oct;36(9):1418-1425. doi: 10.1177/02692163221122325. Epub 2022 Sep 14. PMID 36113084
- [Background] Namisango E, Bristowe K, Murtagh FE, Downing J, Powell RA, Abas M, Lohfeld L, Ali Z, Atieno M, Haufiku D, Guma S, Luyirika EB, Mwangi-Powell FN, Higginson IJ, Harding R. Towards person-centred quality care for children with life-limiting and life-threatening illness: Self-reported symptoms, concerns and priority outcomes from a multi-country qualitative study. Palliat Med. 2020 Mar;34(3):319-335. doi: 10.1177/0269216319900137. Epub 2020 Feb 21. PMID 32081084
- [Background] Coombes LH, Wiseman T, Lucas G, Sangha A, Murtagh FE. Health-related quality-of-life outcome measures in paediatric palliative care: A systematic review of psychometric properties and feasibility of use. Palliat Med. 2016 Dec;30(10):935-949. doi: 10.1177/0269216316649155. Epub 2016 May 31. PMID 27247087
- [Background] Coombes L, Harethardottir D, Braybrook D, Roach A, Scott H, Bristowe K, Ellis-Smith C, Downing J, Bluebond-Langner M, Fraser LK, Murtagh FEM, Harding R. Design and Administration of Patient-Centred Outcome Measures: The Perspectives of Children and Young People with Life-Limiting or Life-Threatening Conditions and Their Family Members. Patient. 2023 Sep;16(5):473-483. doi: 10.1007/s40271-023-00627-w. Epub 2023 May 23. PMID 37221441
- [Background] Scott HM, Coombes L, Braybrook D, Roach A, Harethardottir D, Bristowe K, Ellis-Smith C, Downing J, Murtagh FE, Farsides B, Fraser LK, Bluebond-Langner M, Harding R. Spiritual, religious, and existential concerns of children and young people with life-limiting and life-threatening conditions: A qualitative interview study. Palliat Med. 2023 Jun;37(6):856-865. doi: 10.1177/02692163231165101. Epub 2023 Mar 28. PMID 36978266
- [Background] Coombes L, Braybrook D, Roach A, Scott H, Harethardottir D, Bristowe K, Ellis-Smith C, Bluebond-Langner M, Fraser LK, Downing J, Farsides B, Murtagh FEM, Harding R; C-POS. Achieving child-centred care for children and young people with life-limiting and life-threatening conditions-a qualitative interview study. Eur J Pediatr. 2022 Oct;181(10):3739-3752. doi: 10.1007/s00431-022-04566-w. Epub 2022 Aug 12. PMID 35953678
- [Background] McLorie EV, Hackett J, Fraser LK. Understanding parents' experiences of care for children with medical complexity in England: a qualitative study. BMJ Paediatr Open. 2023 Aug;7(1):e002057. doi: 10.1136/bmjpo-2023-002057. PMID 37550084
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Roach A, Braybrook D, Marshall S. Reflective insights from developing a palliative care children and young people's advisory group. Palliat Med. 2021 Mar;35(3):621-624. doi: 10.1177/0269216320976035. Epub 2021 Jan 12. PMID 33435853
- [Background] Coghlan, A.T., Preskill, H., and Tzavaras Catsambas, T. (2003). An overview of appreciative inquiry in evaluation. New Directions for Evaluation 2003(100), 5-22.
- [Background] Cohen E, Bruce-Barrett C, Kingsnorth S, Keilty K, Cooper A, Daub S. Integrated complex care model: lessons learned from inter-organizational partnership. Healthc Q. 2011;14 Spec No 3:64-70. doi: 10.12927/hcq.0000.22580. PMID 22008576
- [Background] Kaushik, V., and Walsh, C.A. (2019). Pragmatism as a research paradigm and its implications for social work research. Social Sciences 8(9), 255.
- [Background] Bedendo A, Hinde S, Beresford B, Papworth A, Phillips B, Vasudevan C, McLorie E, Walker G, Peat G, Weatherly H, Feltbower R, Hewitt C, Haynes A, Murtagh F, Noyes J, Hackett J, Hain R, Oddie S, Subramanian G, Fraser L. Consultant-led UK paediatric palliative care services: professional configuration, services, funding. BMJ Support Palliat Care. 2023 Aug 9:spcare-2023-004172. doi: 10.1136/spcare-2023-004172. Online ahead of print. PMID 37558392
- [Background] Coombes L, Bristowe K, Ellis-Smith C, Aworinde J, Fraser LK, Downing J, Bluebond-Langner M, Chambers L, Murtagh FEM, Harding R. Enhancing validity, reliability and participation in self-reported health outcome measurement for children and young people: a systematic review of recall period, response scale format, and administration modality. Qual Life Res. 2021 Jul;30(7):1803-1832. doi: 10.1007/s11136-021-02814-4. Epub 2021 Mar 18. PMID 33738710
- [Background] Coombes L, Harethardottir D, Braybrook D, Scott HM, Bristowe K, Ellis-Smith C, Fraser LK, Downing J, Bluebond-Langner M, Murtagh FE, Harding R. Achieving consensus on priority items for paediatric palliative care outcome measurement: Results from a modified Delphi survey, engagement with a children's research involvement group and expert item generation. Palliat Med. 2023 Dec;37(10):1509-1519. doi: 10.1177/02692163231205126. Epub 2023 Oct 18. PMID 37853579
- [Background] Murtagh FEM, Guo P, Firth A, Yip KM, Ramsenthaler C, Douiri A, Pinto C, Pask S, Dzingina M, Davies JM, O'Brien S, Edwards B, Groeneveld EI, Hocaoglu M, Bausewein C, Higginson IJ. A casemix classification for those receiving specialist palliative care during their last year of life across England: the C-CHANGE research programme. Southampton (UK): National Institute for Health and Care Research; 2023 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK597740/ PMID 38048413
- [Background] Pask S, Pinto C, Bristowe K, van Vliet L, Nicholson C, Evans CJ, George R, Bailey K, Davies JM, Guo P, Daveson BA, Higginson IJ, Murtagh FEM. A framework for complexity in palliative care: A qualitative study with patients, family carers and professionals. Palliat Med. 2018 Jun;32(6):1078-1090. doi: 10.1177/0269216318757622. Epub 2018 Feb 19. No abstract available. PMID 29457743
- [Background] Cassidy L, Quirke MB, Alexander D, Greene J, Hill K, Connolly M, Brenner M. Integrated care for children living with complex care needs: an evolutionary concept analysis. Eur J Pediatr. 2023 Apr;182(4):1517-1532. doi: 10.1007/s00431-023-04851-2. Epub 2023 Feb 13. PMID 36780041
- [Background] Hain R, Devins M, Hastings R, Noyes J. Paediatric palliative care: development and pilot study of a 'Directory' of life-limiting conditions. BMC Palliat Care. 2013 Dec 11;12(1):43. doi: 10.1186/1472-684X-12-43. PMID 24330676
- [Background] Horridge KA, Harvey C, McGarry K, Williams J, Whitlingum G, Busk M, Fox S, Baird G, Spencer A. Quantifying multifaceted needs captured at the point of care. Development of a Disabilities Terminology Set and Disabilities Complexity Scale. Dev Med Child Neurol. 2016 Jun;58(6):570-80. doi: 10.1111/dmcn.13102. Epub 2016 Mar 23. PMID 27009933
- [Background] Royal College of Paediatrics and Child Health. (2021). Our vision for the future of paediatrics in the UK: Executive Summary. Royal College of Paediatrics and Child Health
- [Background] Cohen E, Kuo DZ, Agrawal R, Berry JG, Bhagat SK, Simon TD, Srivastava R. Children with medical complexity: an emerging population for clinical and research initiatives. Pediatrics. 2011 Mar;127(3):529-38. doi: 10.1542/peds.2010-0910. Epub 2011 Feb 21. PMID 21339266
- [Background] Jemal, J., and Kenley, A. (2023). Wasting Money, Wasting potential - the costs of SEND tribunals. Pro Bono Economics
- [Background] Ahmedzai SH. Legal right to palliative care wouldn't be needed if the hospice movement didn't operate outside the NHS. BMJ. 2022 Jun 16;377:o1422. doi: 10.1136/bmj.o1422. No abstract available. PMID 35710112
- [Background] Fisher V, Atkin K, Ewing G, Grande G, Fraser LK. Assessing the suitability of the Carer Support Needs Assessment Tool (CSNAT-Paediatric) for use with parents of children with a life-limiting condition: A qualitative secondary analysis. Palliat Med. 2024 Jan;38(1):100-109. doi: 10.1177/02692163231214471. Epub 2023 Dec 23. PMID 38142279
- [Background] Pinney, A. (2017). Understanding the needs of disabled children with complex needs or life-limiting conditions: What can we learn from national data? Council for disabled children, The True Colours Trust
- [Background] Page BF, Hinton L, Harrop E, Vincent C. The challenges of caring for children who require complex medical care at home: 'The go between for everyone is the parent and as the parent that's an awful lot of responsibility'. Health Expect. 2020 Oct;23(5):1144-1154. doi: 10.1111/hex.13092. Epub 2020 Jun 16. PMID 32542954
- [Background] Fraser LK, Parslow R. Children with life-limiting conditions in paediatric intensive care units: a national cohort, data linkage study. Arch Dis Child. 2018 Jun;103(6):540-547. doi: 10.1136/archdischild-2017-312638. Epub 2017 Jul 13. PMID 28705790
- [Background] Fraser LK, Gibson-Smith D, Jarvis S, Norman P, Parslow RC. Estimating the current and future prevalence of life-limiting conditions in children in England. Palliat Med. 2021 Oct;35(9):1641-1651. doi: 10.1177/0269216320975308. Epub 2020 Dec 15. PMID 33323043
- [Background] Fraser LK, Miller M, Hain R, Norman P, Aldridge J, McKinney PA, Parslow RC. Rising national prevalence of life-limiting conditions in children in England. Pediatrics. 2012 Apr;129(4):e923-9. doi: 10.1542/peds.2011-2846. Epub 2012 Mar 12. PMID 22412035
- [Background] Chambers, L. (2018). A Guide to Children's Palliative Care: Supporting babies, children and young people with life-limiting and life-threatening conditions and their families. Together for Short Lives
- See also: The CoLab Partnership — https://www.colabpartnership.org.uk
- See also: PROSPERO Registration: A realist review of multisectoral integrated care for children and young people with medical complexity. — https://www.crd.york.ac.uk/PROSPERO/view/CRD420250653996
- See also: UK Standards for Public Involvement — https://sites.google.com/nihr.ac.uk/pi-standards/home
- See also: Difference between children's and adult palliative care.[online]. (Together for Short Lives — https://www.togetherforshortlives.org.uk/changing-lives/supporting-care-professionals/introduction-childrens-palliative-care
- See also: Hope House Children's Hospices — https://www.hopehouse.org.uk/trends-report